## Tailored Self-Management of TMD Pain using Health Information Technology

**NIDCR Protocol Number: 16-054-E** 

NIDCR Grant Number: U01 DE025609

Principal Investigator: James Fricton, DDS, MS

March 20, 2017

## **Final Analysis Plan**

We will perform the following analysis and present results in preparation of the full study. The Primary outcomes for this study are acceptability and feasibility of the methods. The study is not sufficiently powered to test for mean changes from baseline to follow-up. Thus, we will conduct the following descriptive analysis at noted in the outcome measures:

- Number of participants, baseline characteristics and outcomes at baseline will be summarized descriptively
- Summary measures will include mean values (standard deviation SD) for continuous variables and frequency distribution for categorical variables.
- Outcome measures will be analyzed for departure of normality, and standard transformations will be applied.
- Percent of participants completing the measures for outcomes, mediating and moderating factors at baseline and each follow-up periods

The acceptability of the outcomes, mediating and moderating measures at baseline and followup periods